CLINICAL TRIAL: NCT07359482
Title: sElective Serotonin reuPtake inhibitoRs In posT-covid: ESPRIT
Brief Title: sElective Serotonin reuPtake inhibitoRs In posT-covid
Acronym: ESPRIT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Pythia Nieuwkerk, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-519540-32-00; 11080022420014 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post-COVID; POST-Covid 19; Post-COVID Conditions
Keywords: post-COVID; fluvoxamine; fatigue; biomarkers
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue | interventions — Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Two arm study in which post-COVID patients are randomly assigned to fluvoxamine or placebo in a double blind way.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Fluvoxamine.
  Interventions: Drug: Fluvoxamine
- Control arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine — Subject are randomized in a double-blind manner (1:1 ratio) between fluvoxamine and placebo. During the first week subjects will receive a low dose daily dose of fluvoxamine of 25 mg or placebo. In the second week, subjects will receive a daily dose of 50 mg or placebo. From week 3 onwards, the fluvoxamine or placebo dose is increased by daily 50 mg every 6 days in a blinded manner but will not be further increased if participants are unwilling to accept a dose increase. For doses higher than 100 mg per day, dosing is done twice daily. The dose is increased to a maximum of 200 mg per day (i.e. 100 mg bid). The minimal daily dose is 50 mg.
  Arms: Intervention arm
Drug: Placebo — Subject are randomized in a double-blind manner (1:1 ratio) between fluvoxamine and placebo. During the first week subjects will receive a low dose daily dose of fluvoxamine of 25 mg or placebo. In the second week, subjects will receive a daily dose of 50 mg or placebo. From week 3 onwards, the fluvoxamine or placebo dose is increased by daily 50 mg every 6 days in a blinded manner but will not be further increased if participants are unwilling to accept a dose increase. For doses higher than 100 mg per day, dosing is done twice daily. The dose is increased to a maximum of 200 mg per day (i.e. 100 mg bid). The minimal daily dose is 50 mg.
  Arms: Control arm

SUMMARY:
Fatigue, cognitive problems, post-exertional malaise (PEM) and postural orthostatic tachycardia syndrome (POTS) are common and debilitating symptoms after COVID-19. The pathophysiology of post-COVID is not well understood and there is no established biomedical treatment. Treatment options for post-COVID are thus much needed.

A promising candidate intervention is fluvoxamine, a selective serotonin reuptake inhibitor (SSRI), that may reduce post-COVID symptoms because of its regulatory effect on the (neuro) immune system, the hypothalamic-pituitary-adrenal (HPA) axis and the tryptophan system. We will randomize 160 participants to either fluvoxamine or placebo for 12 weeks.

We will use advanced functional neuroimaging techniques during cognitive challenge (optional substudy) and plasma biomarkers (inflammatory markers, cortisol, serotonin, IDO-2 activity), to facilitate identifying potential mechanistic pathways of post -COVID treatment.

DETAILED DESCRIPTION:
In this randomized placebo-controlled trial, we will investigate the effectiveness of fluvoxamine in reducing fatigue severity (primary outcome), cognitive problems, PEM and POTS after 12 weeks of treatment in 160 post-COVID patients.

Moreover, we will study treatment-emergent changes in plasma biomarkers, including blood-based neuro)inflammatory markers, cortisol, serotonin, aryl hydrocarbon receptor -indoleamine 2,3-dioxygenase-2 (IDO-2) and kynurenine pathway (KP) metabolites for potential mechanistic pathways of post-COVID treatment.

Numerous studies have indicated involvement of brain dysfunction in post COVID, which also relate to the degree of symptom severity (e.g. fatigue / cognitive problems). In an optional neuro-imaging sub-study, we will use functional neuroimaging techniques with and without cognitive challenge to gain a better understanding of the brain functioning and structure in long COVID during fluvoxamine treatment versus placebo.

Objectives:

* To determine if fluvoxamine treatment (50 mg to 200 mg daily dosing) results in lower levels of fatigue severity than placebo after 12 weeks of treatment (primary).
* To determine if fluvoxamine treatment results in lower levels of PEM and POTS and a better cognitive functioning and health-related quality of life (HRQL) than placebo.
* To determine if changes in symptoms, i.e. fatigue severity, PEM, POTS, cognitive symptoms, are related to changes in biomarkers, i.e., (neuro)inflammation markers, cortisol, serotonin and IDO-2 -KP metabolites.
* To determine if biomarkers, i.e., (neuro)inflammation markers, cortisol, serotonin and IDO-2- KP metabolites, change from baseline to week 12 in participants who received fluvoxamine.

Optional Neuro-imaging sub-study:

-To determine which changes occur on functional brain imaging, brain metabolites and neuroinflammation during cognitive challenge and to determine if this brain response to cognitive challenge changes after fluvoxamine treatment versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years
* Severely fatigued (CIS fatigue score ≥ 35) at screening
* Fatigue started/increased significantly after Covid-19 (self-declared)
* Fatigue symptoms must be present for at least 3 months following the acute infection.
* Self-reported confirmation of having a SARS-CoV-2 infection by: Positive SARS-CoV-2 nucleic acid amplification test (NAAT), such as PCR; Positive SARS-CoV-2 rapid diagnostic test, including home-administered tests; COVID-19 diagnosis by a medical specialist (GP or in-hospital), based on the above or other clinical test or assessments. The above information will not be verified in medical records.
* Command of Dutch or English language to complete questionnaires
* Able to participate in video calling.
* Willing and able to provide informed consent
* Allowing the trial team to exchange medical information that is relevant for the participants' safety and trial assessments with their GP and pharmacy.

Exclusion Criteria:

* Use of medication with interaction with fluvoxamine that cannot be discontinued
* Hospitalized in the acute phase of Covid-19
* Psychiatric/somatic disorders that could explain the severity of fatigue
* Neurodegenerative disorders (i.e. M Parkinson, Multiple sclerosis, M Alzheimer)
* Suicidality (current or recent) (according to WHO suicide screener)
* Starting or started with other medication intended to reduce post-covid symptoms during the last 2 months
* Pregnancy (a positive urine or serum pregnancy test) or unwilling to use standard contraception
* Brugada- or Long QT interval syndrome
* epilepsy, porphyria, history of severe liver impairment
* known allergies to fluvoxamine or placebo/excipients
* known current alcohol or drug use problems.
* Bleeding disorders and past medical history of bleeding gastric or duodenal ulcers or other significant bleeding disorders
* claustrophobia (optional MRI substudy)
* having metal implants (optional MRI substudy)
* inability to lay still for 45 minutes (optional MRI substudy)
* Neurotrauma/ large stroke or brain abnormalities interfering with image analyses (optional MRI substudy)
* Inability to come to the Amsterdam UMC (optional MRI substudy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity | week 12
  fatigue score CIS-20R

SECONDARY OUTCOMES:
Fatigue severity | week 4, 8, 12
  PROMIS fatigue 8
Cognitive functioning | week 4, 8, 12
  PROMIS cognitive function 8a
Cognitive functioning | week 4, 8, 12
  Concentration score CIS-20R
PEM | week 4, 8, 12
  DSQ-PEM
POTS (National Aeronautics and Space Administration (NASA) lean test | week 12
  NASA lean test
POTS | week 4, 8, 12
  DSQ-POTS
Health-related Quality of Life | week 4, 8, 12
  PROMIS-29
Disability | week 4, 8, 12
  Bell disability score
Side effects | week 12
  Antidepressant Side Effect Checklist-21 (ASEC-21)
Side effects | week 12
  Frequency, Intensity, Burden of Side Effects Rating scale (FIBSER scale)
Brain Perfusion (optional MRI substudy) | week 12
  Arterial Spin Labeling
Brain functioning and connectivity (optional MRI substudy) | week 12
  During resting-state and cognitive effort (challenging N-back (3-back vs. 0-back) on functional MRI
Brain metabolites and neuroinflammation (optional MRI substudy) | week 12
  Magnetic Resonance Spectroscopy

OTHER OUTCOMES:
Biomarkers | week 12
  (neuro) inflammation markers, corticoid receptor activity and cortisol, serotonin, IDO-2/ KP metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Sharing will be in accordance with Dutch privacy laws and regulations.
Supporting Information: Study Protocol, SAP, ICF